CLINICAL TRIAL: NCT02385656
Title: The Efficacy and Tolerability of Modafinil for Fatigue and Daytime Sleepiness in Cancer Patients: Preliminary Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, In-Young Yoon, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-1302/191-003
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): Subjects who take modafinil for cancer-related fatigue for 4 weeks.
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — 200mg of modafinil daily for 4 weeks
  Other Names: Provigil

SUMMARY:
Open-pilot study for the efficacy and tolerability of modafinil on the fatigue and somnolence in cancer-patients.

DETAILED DESCRIPTION:
This is an open-pilot study for the efficacy and tolerability of modafinil on the fatigue and somnolence in cancer-patients. Patients with moderate to severe cancer-related fatigue will be treated with modafinil for 4 weeks and psychological tests including self-questionnaire, cognitive test, sleep-wake cycle, quantitative electroencephalogram(QEEG) will be applied pre- and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* solid cancer patient
* age of 20-65 years old
* subjects who scored =4 or >4 on the Brief Fatigue Inventory
* subjects with informed consent

Exclusion Criteria:

* metastatic cancer(stage IV)
* with psychotic symptoms such as delusion and hallucination or with suicidal risk
* with delirium or dementia
* current medication of cognitive enhancer or psychostimulant uncontrolled medical illness
* current medications that are contraindicated or not recommended for co-administration with modafinil

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
severity of fatigue (Brief Fatigue Inventory) | 4 weeks
  Brief Fatigue Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Inyoung Yoon, M.D., Ph.D., Principal Investigator — Department of Psychiatry, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea